CLINICAL TRIAL: NCT03756597
Title: PAN-study: Pan-Cancer Early Detection Study
Brief Title: PAN-study: Pan-Cancer Early Detection Study (PAN)
Status: Completed | Type: Observational
Sponsor: Owlstone Ltd (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: PAN
Record Dates: First submitted 2018-10-16; First posted 2018-11-28 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer; Esophageal Cancer; Liver Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients will inhale room air from which environmental VOCs have been removed to prevent contamination of the sample. The mask contains a CO2 sensor that drives two micro-pumps in the mask that sample alveolar and bronchial breath separately. This is relevant because different cancer biomarkers can be found in different portions of breath. During the procedure the breath will automatically be sampled onto four sorbent tubes to collect a total of 1.5L of breath. The procedure will normally take around 10 minutes, very rarely exceeding 15 minutes if exhaled volumes are small. After collection, the sorbent tubes are stored in the refrigerator at 4-8°C until shipment to Owlstone Medical. For those participating in the washout sub study, up to 6 samples will be obtained at various timepoints in one day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cases Pathway A: Case pathway A - Intention to diagnose population
  Only patients with a very high clinical suspicion based on imaging are scheduled for surgical procedures.Subjects with a confirmed diagnosis of cancer after clinical work-up will be labelled cases. of the study.
  Patients with Gastric or Oesophageal cancer will be recruited after confirmation of their diagnosis but prior to initiation of therapy.
  Interventions: Device: ReCIVA; Device: CASPER
- Clinical Controls: Clinical controls represent subjects that:
  * Are suspected of the same cancer or part of an at risk-group
  * Have undergone full per-guideline diagnostic work-up, resulting in confirmation the subject does not have cancer (see section 6)
  * Is matched to the case for age, gender and known risk-factors specific to that tumour type (section 5.4)
  Interventions: Device: ReCIVA; Device: CASPER
- Healthy volunteers: Healthy volunteers will be recruited from the clinical research facility at Addenbrooke's Hospital (Cambridge) or from the Cambridge BioResource. These subjects will be selected to have a similar age and sex distribution as the overall PAN-study cases.
  Interventions: Device: ReCIVA; Device: CASPER
- Substudy Cases: Patients with a confirmed diagnosis of cirrhosis and providing up to 6 samples will be labelled as the washout substudy cases
  Interventions: Device: ReCIVA; Device: CASPER
- Cases Pathway B: Case pathway B - Confirmed malignancy population
  Patients with a Gastric, Liver or Oesophageal cancer will be recruited after confirmation of their diagnosis but prior to initiation of therapy. Patients will be recruited by research staff at the clinic they are referred to for diagnosis and/or treatment
  Interventions: Device: ReCIVA; Device: CASPER

INTERVENTIONS:
Device: ReCIVA — The ReCIVA breath sampler contains a CO2 and pressure sensor, which allows the operator to monitor the breath sampling procedure and patient comfort. Both the operator and the patient can pause or abort the breath sampling procedure within seconds by removing the mask. The time investment required from patients is approximately 15 minutes for consenting and medical history and 10 minutes per breath collection.
Device: CASPER — Minimizes contamination of breath samples by external VOCs Removes need for clean air supply line

SUMMARY:
The PAN-cancer Early Detection study or PAN-study is a prospective cross-sectional observational case-control study evaluating whether Breath Biopsy can differentiate between patients with and without different cancer types by comparing breath biomarkers for a range of cancer types including patients with gastric, oesophageal, and liver cancer.

The research may be extended to include also pancreatic, renal, prostate and bladder cancer patients, however in agreement between Cambridge University Hospital NHS Foundation Trust, University of Cambridge, CRUK and Owlstone Medical recruitment in these arms will not start until further notice. When recruitment is planned to start in these arms, Owlstone Medical will ensure to notify the REC. Subjects with a histologically confirmed cancer will be recruited from CUH by local research staff. Breath samples will be collected by means of the ReCIVA breath sampler which requires tidal breathing into a face mask for around 10 minutes. A cancer free control subject matched for age, sex and tumour specific risk factors will be recruited and sampled.

DETAILED DESCRIPTION:
There is a pressing need for techniques that allow detection of cancer at an earlier stage when curative treatment is more likely. Exhaled biomarkers are known to reflect a wide range of metabolic processes, including those related to cancer such as the Warburg effect. Owlstone Medical Ltd (hereafter referred to as Owlstone Medical) has developed Breath Biopsy; a workflow to collect and analyse breath Volatile Organic Compounds (VOCs) in a highly standardised way. The PAN-study is a collaborative effort between Cambridge University Hospitals NHS Foundation Trust (CUH), University of Cambridge (UoC), Cancer Research United Kingdom (CRUK) and Owlstone Medical to evaluate the potential of Breath Biopsy to detect various types of cancer by profiling breath metabolites.

The PAN-cancer Early Detection study or PAN-study is a prospective cross-sectional observational case-control study evaluating whether Breath Biopsy can differentiate between patients with and without different cancer types by comparing breath biomarkers for a range of cancer types including patients with gastric, oesophageal, and liver cancer.

The research may be extended to include also pancreatic, renal, prostate and bladder cancer patients, however in agreement between Cambridge University Hospital NHS Foundation Trust, University of Cambridge, CRUK and Owlstone Medical recruitment in these arms will not start until further notice. When recruitment is planned to start in these arms, Owlstone Medical will ensure to notify the REC. Subjects with a histologically confirmed cancer will be recruited from CUH by local research staff. Breath samples will be collected by means of the ReCIVA breath sampler which requires tidal breathing into a face mask for around 10 minutes. A cancer free control subject matched for age, sex and tumour specific risk factors will be recruited and sampled. Breath samples will be shipped to Owlstone Medical for analysis of breath biomarkers by Gas Chromatography-Time Of Flight-Mass Spectrometry (GC-TOF-MS) and Gas Chromatography-Field Asymmetric Ion Mobility Spectrometry (GC-FAIMS).

This study will be the first step towards evaluating VOCs analysis as a test to improve early detection rates for cancer with future applicability to primary care. Ultimately, such a research program could enable low cost and widespread targeted screening programs for cancer.

In a subset of up to 12 patients with cirrhosis and 12 healthy volunteers, a sub study will be conducted to measure the washout of limonene after ingestion of a standardised quantity of limonene under controlled circumstance for food and drink intake.

The objective of this limonene sub-study is to demonstrate that limonene is a biomarker that differentiates between healthy individuals and cirrhotic patients with Child-Pugh grade A and B with or without HCC as a comorbidity.

Participants will be asked to visit the clinical site to provide 6 breath samples at different timepoints before and after ingestion of limonene. Participants will be asked to fast overnight for 10 hours, not to have brushed their teeth for 2 hours prior to first breath sample and not be a current smoker or should not have smoked in the past 6 months. Non-abstinent patients with alcohol related liver disease or participants who drink to excess daily will be excluded from this sub-study.

ELIGIBILITY:
5.1. General inclusion criteria

1. Aged 30 years or over
2. Ability to provide informed consent

5.2. General exclusion criteria

1. (Anticipated) inability to complete the breath sampling procedure due to e.g. inability to maintain adequate ventilation unaided or claustrophobia
2. Participation in a Clinical Trial Investigational Medicinal Product (CTIMP) during the 28 days prior to breath biopsy.
3. Any biopsy or endoscopic procedure conducted during the past 48 hours. A breath sample can be collected >48 hours post procedure.
4. Any disorder that is not stable in the opinion of the investigator. Specifically, subjects should be excluded if:

   4.1. Currently in the process of investigation for a malignancy other than the tumours of interest to this study.

   4.2. A history of malignancy, unless treated with curative intent and cancer-free at least 2 years prior to inclusion. Patients previously treated for highly localised disease e.g. basal cell carcinoma, localised squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that curative therapy was completed at least 12 months prior to inclusion.

   4.3. A history of the malignancy the patient is currently being investigated for. E.g. a patient suspected of gastric cancer with previous gastric cancer in medical history 4.4. Known active bacterial, fungal or viral infection including but not limited to upper respiratory tract infection, tuberculosis, pneumonia, cystitis, pyelonephritis, gastritis, prostatitis or viral hepatitis. Patients can be recruited after being symptom free for at least 2 weeks for mild infections and 6 weeks if admitted to the hospital and/or treated with i.v. antibiotics.

   4.5. Documented history of a clinically important lung condition other than asthma or COPD e.g., active lung infection, , bronchiectasis, cystic fibrosis, primary ciliary dyskinesia, allergic bronchopulmonary aspergillosis/mycosis, pulmonary fibrosis or hypersensitivity pneumonitis, α1- antitrypsin deficiency. If α1- antitrypsin deficiency is diagnosed after a breath sample has been taken, the patient sample may still be used for analysis. α1- antitrypsin carriers are eligible for the study.

   4.6. Asthma or COPD exacerbation requiring hospitalisation and/or administration of oral prednisolone in past 6 weeks.

   4.7. Renal failure stages 3b and above (eGFR 45ml/min or less) 4.8. Any hospitalisation for symptoms unrelated to the clinical presentation of the tumour under investigation during the past 6 weeks.
5. Immunocompromised patients: specifically, patients with Acquired Immune Deficiency Syndrome (AIDS) (HIV with normal blood counts is eligible), inborn or acquired severe immune-deficiency including those caused by pharmacological treatment.
6. Documented history of pulmonary surgery or endobronchial interventional procedures other than biopsy, lavage or bronchial brushings. These include surgical resection, VATS, bronchial thermoplasty and coiling.
7. Applicable for the limonene sub-study only (see section 4.1): Non-abstinent participants with alcohol related liver disease or participants who drink to excess daily.
8. Applicable for the limonene sub-study only (see section 4.1): Current smokers (or e-cigarette users) or participants who have smoked (or used e-cigarettes) in the past 6 months prior to baseline sample.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion and exclusion criteria for the various study populations are detailed above. General inclusion and exclusion criteria which apply to all study subjects are detailed followed by indication specific criteria are also detailed for both inclusion and exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Primary endpoints; accuracy of breath biopsy to discriminate between individuals with and without cancer | 3 years
  o These will include gastric, oesophageal and liver and matched controls. This analysis will be conducted by combining cases and matched controls across all cancer types as well as when stratified per tumour type. If supported by literature on the presence of potential biomarkers related to pancreatic, renal, prostate, and bladder tumours similar analysis will be done in samples collected in patients diagnosed with these cancer types and controls.

SECONDARY OUTCOMES:
Patient feedback on usability and acceptability of Breath Biopsy as assessed using a a structured interview | 3 years
  * Patient feedback on usability and acceptability, including willingness to participate.
  * Qualitative review of barriers to adoption for study subjects and health professionals.

OTHER OUTCOMES:
Exploratory endpoints; influence of tumour phenotype on breath VOCs: | 3 years
  * Comparison between exhaled breath VOCs of different tumour types.
  * Impact of tumour stage, pre-cancerous condition and benign tumours on VOC levels.
  * Performance of breath test relative to and in combination with epidemiological risk models.

CONTACTS AND LOCATIONS:
Overall Officials: Marc P van der Schee, MD, PhD, Study Director — +01223 428200; Prof Rebecca Fitzgerald, MD, PhD, Study Chair — Cambridge University Hospital; Massimiliano di Pietro, MD, PhD, Principal Investigator — Cambridge University Hospital; Mr Vincent J Gnanapragasam, MD, PhD, Principal Investigator — Cambridge University Hospital; Mr Grant Stewart, MD, PhD, Principal Investigator — Cambridge University Hospital; Dr Godfrey Edmund, MD, PhD, Principal Investigator — Cambridge University Hospital; Miss Alexandra Colquhoun,, Principal Investigator — Cambridge University Hospital; Dr Victoria Snowdon, Principal Investigator — Cambridge University Hospital; Dr Matthew Hoare, Principal Investigator — Cambridge University Hospital; Dr Michael Allison, Principal Investigator — Cambridge University Hospital
Locations (1):
- Cambridge University Hospital NHS, Cambridge, United Kingdom

REFERENCES:
- See also: PAN study website — https://www.owlstonemedical.com/clinical-pipeline/pan/